CLINICAL TRIAL: NCT05368428
Title: Single-Institution Trial Investigating the Effectiveness of Transcutaneous Electrical Nerve Stimulation (TENS) in Taxane Induced Peripheral Neuropathy (CIPN) in Patients With Early Stage Breast Cancer
Brief Title: Transcutaneous Electrical Nerve Stimulation in Chemotherapy Induced Peripheral Neuropathy in Patients With Stage I-III Early Stage Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Manali Bhave, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00003705; NCI-2022-01726 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00003705 (Other: Emory University Hospital/Winship Cancer Institute); WINSHIP5501-21 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Chemotherapy-Induced Peripheral Neuropathy; Early Stage Breast Carcinoma; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (TENS) (Experimental): Patients undergo TENS therapy daily over 1 hour for 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Other: Transcutaneous Electrical Nerve Stimulation — Undergo TENS
  Other Names: TENS; transcutaneous electric nerve stimulation

SUMMARY:
This phase II trial examines transcutaneous electrical nerve stimulation (TENS) in patients with stage I-III breast cancer with chemotherapy induced peripheral neuropathy. TENS is a procedure in which mild electric currents are applied to some areas of the skin to potentially improve neuropathy. This trial may help determine if TENS is feasible and effective for the treatment of peripheral neuropathy symptoms while on chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the feasibility of daily transcutaneous electrical nerve stimulation (TENS) by measuring participant adherence to TENS for two weeks.

SECONDARY OBJECTIVES:

I. To evaluate the change in patient reported outcome (PRO) measures of symptoms (e.g. pain, tingling, numbness) and functional impairment.

II. To evaluate the change in objective measures of neuropathy over the study period through bedside monofilament testing.

TERTIARY/EXPLORATORY OBJECTIVES:

I. To collect data on the type and use frequency of non-TENS chemotherapy-induced peripheral neuropathy (CIPN) treatments (e.g. neuropathic agents and doses) both at baseline and over the duration of the trial (six weeks).

II. To measure the number of chemotherapy dose-limiting events (dose reductions, delays, discontinuations) over the duration of the trial.

OUTLINE:

Patients undergo TENS therapy at home daily over 1 hour for 14 days in the absence of unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven stage I-III breast cancer actively undergoing neoadjuvant or adjuvant chemotherapy regimen that contains paclitaxel or docetaxel.
* At least Common Terminology Criteria for Adverse Events (CTCAE) grade 1 CIPN in hands or feet attributed to taxane chemotherapy.
* Actively undergoing paclitaxel or docetaxel with plans to continue during the two-week TENS treatment.
* Age >= 18 years
* For females of child-bearing potential, negative serum or urine pregnancy test within 14 days prior to starting TENS
* Given the potential concern that TENS could induce uterine contractions or interfere with fetal cardiac conduction, female of child-bearing potential (FCBP) must have a negative serum or urine pregnancy test prior to starting therapy
* Female of childbearing potential (FCBP) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of TENS treatment. Should a woman become pregnant or suspect she is pregnant during the two weeks of TENS, she should inform her treating physician immediately. A female of childbearing potential (FCBP) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Willingness and ability of the subject to comply with scheduled visits, TENS administration plan, other study procedures, and study restrictions.
* Evidence of a personally signed informed consent indicating that the subject has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential risks and discomforts, potential benefits, and other pertinent aspects of study participation
* Patients must have the psychological ability and general health that permits completion of the study requirements and required follow up
* Women of child bearing potential (FCBP) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Skin wounds, skin breakdown or edema at the site of TENS electrode pad placement
* History of epilepsy
* Implanted electronic device including a cardiac pacemaker, defibrillator, pain pump etc.
* Pre-existing neuropathy
* Prior exposure to neurotoxic chemotherapy
* Previous use of TENS for CIPN
* Prisoners or an adult who is unable to consent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2026-01-23 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the Feasibility of Daily TENS by Measuring Participant Adherence to TENS for Two Weeks | Up to 2 weeks
  Adherence for each trial participant will be calculated by summing the number of one-hour TENS sessions completed and dividing by 14 total treatments. Adherence for the cohort will be summarized descriptively using descriptive statistics.

SECONDARY OUTCOMES:
Change in Patient Reported Outcomes Measurement Information System 29 score | At baseline and 2 and 6 weeks
  Change in Patient Reported Outcomes Measurement Information System 29 score at two and six weeks compared to baseline
  * Physical Function scored on a scale from "without any difficulty" (maximum value) to "unable to do" (minimum value)
  * Anxiety scored on a scale from "always" (maximum value) to "never" (minimum value)
  * Depression scored on a scale from "always"(maximum value) to "never" (minimum value)
  * Fatigue scored on a scale of "very much" (maximum value) to "not at all" (minimum value)
  * Sleep Disturbance scored on a scale from "very good" (maximum value) to "very poor" (minimum value)
  * Ability to Participate in Social Roles and Activities" scored on a scale from "never" (maximum value) to "always" (minimum value)
  * Pain Interference scored on a scale from "very much" (maximum value) to "not at all" (minimum value)
  * Pain Intensity scored on a scale of 0-10, where "10" is the maximum value and "0" is the minimum value.
Change in Monofilament Testing | At baseline and 2 and 6 weeks
  Testing at two and six weeks compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Manali Bhave, MD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (3):
- United States (3):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia